CLINICAL TRIAL: NCT02657395
Title: PriMatrix Utilization to Achieve Dental Root Coverage
Brief Title: Root Coverage Using a Xenograph for Treatment of Gingival Recession
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Daniel Assad, Consultant, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15-006568
Record Dates: First submitted 2015-12-16; First posted 2016-01-15 (Estimated); Last update posted 2017-07-25 (Actual); Status verified 2017-07

CONDITIONS: Localized Gingival Recession

STUDY DESIGN:
Intervention Model Description: Bovine collagen matrix -PriMatrix
Oversight: Data Monitoring Committee: No

ARMS (1):
- PriMatrix (Experimental): Use of PriMatrix as a substitute for a subepithelial connective tissue graft under a coronal positioned flap for root coverage.
  Interventions: Device: PriMatrix

INTERVENTIONS:
Device: PriMatrix — Use of PriMatrix under a coronal positioned flap to obtain root coverage.

SUMMARY:
Can a fetal bovine derived membrane serve as an alternative to autogenous tissue for dental root coverage procedures.

DETAILED DESCRIPTION:
PriMatrix (TEI Medical Inc) is a promising collagen membrane derived from fetal bovine dermis. The acellular porous structure of the membrane permits rapid re-vascularization and cellular re-population. The membrane contains a high proportion of type III collagen. Type III collagen helps regulate tissue healing by promoting neoepithelialization and angiogenesis. Wounds grafted with PriMatrix exhibited significantly faster healing rates compared to control wounds while having a minimal foreign body response and early repopulation by progenitor cells.

The ability of PriMatrix to permit neovascularization, reepithelialization, minimal immune response, and population by progenitor cells suggests that it may serve as an ideal alternative to CTG under CPF for root coverage. In this regard, the current study aims to serve as a pilot to test the feasibility of the use of PriMatrix as a graft material under a CPF to attain root coverage of Miller Class I & II defects.

ELIGIBILITY:
* Inclusion Criteria:

  * Adults 18-90 years of age
  * Miller Class I & II defects on maxillary or mandibular teeth
  * At least 1 adjacent non-involved tooth on either side of the included recession defects
  * Keratinized tissue width of ≥2.0 mm
  * Periodontal probing depths of 3 mm or on included teeth
  * Plaque index of 2 or less
  * Bleeding on probing at 30% or less sites
  * Current non-smoker
  * No active infected wounds
* Exclusion Criteria

  * Patients less than 18 years of age
  * Miller Class III, or IV mucogingival defects
  * Miller Class I & II defects without adjacent non-involved teeth
  * CEJ not identifiable
  * Root surface restoration at the defect site
  * Periodontal probing depths greater than 3 mm
  * Plaque index of 2 or greater
  * Bleeding on probing at more than 30% of sites
  * Uncontrolled oral disease
  * Moderate to severe generalized chronic or aggressive periodontitis
  * Oral manifestations of a systemic disease
  * History of previous root coverage procedure, graft, or GTR
  * Current smoker or other tobacco use
  * Alcohol abuse problems
  * Traumatic occlusion impinging on the recession defect
  * Use of intraoral appliances that impinge on the recession defect
  * Intra-oral piercings that impinge on the included defect
  * Uncontrolled systemic health conditions
  * Debilitating systemic or infectious disease
  * Diabetes
  * Heart Disease
  * Uncontrolled heart disease
  * Delayed wound healing
  * Immunocompromised status due to medication or immune system dysfunction
  * Active infection or non-healing wounds
  * Currently pregnant or lactating
  * Long-term steroid use

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2015-10; Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Complete Root Coverage | 6-months
  The percentage of sites showing complete root coverage will be calculated as a percent of treated defects with the marginal gingival located at or above the cement-enamel junction compared to the total defects treated.

SECONDARY OUTCOMES:
Clinical Periodontal Parameters | Baseline, 6-weeks, 4-months, and 6-months
  Determine keratinized tissue width of the augmented region using a UNC-15 mm periodontal probe.
Clinical Periodontal Parameters | Baseline, 6-weeks, 4-months, and 6-months
  Determine periodontal probing depths of the augmented region using a UNC-15 mm periodontal probe.
Clinical Periodontal Parameters | Baseline, 6-weeks, 4-months, and 6-months
  Determine tissue thickness of the augmented region using a UNC-15 mm periodontal probe.
Clinical Periodontal Parameters | Baseline, 6-weeks, 4-months, and 6-months
  Determine clinical attachment levels of the augmented region using a UNC-15 mm periodontal probe.
Pain Levels | 1-week, 2-weeks, 4-weeks, and 6-months
  Visual analog scale questionnaire will be completed consisting of 5 to 6 questions at each appointment.
Mean Root Coverage Obtained | Baseline, 6-weeks, 4-months, and 6-months
  Percentage of baseline root coverage obtained as a fraction of initial recession depth will be measured using a UNC-15 mm periodontal probe.
Gingival Health | Baseline, 6-weeks, 4-months, and 6-months
  Gingival health will be evaluated visually using Silness and Loe Gingival index.
Plaque Levels | Baseline, 6-weeks, 4-months, and 6-months
  Plaque levels will be evaluated using the Quigley and Hein plaque index.
Esthetic Outcomes | 1-week, 2-weeks, 4-weeks, and 6-months
  Visual analog scale questionnaire will be completed consisting of 5 to 6 questions at each appointment.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Assad, DDS, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Undecided